CLINICAL TRIAL: NCT01682993
Title: Topography Guided Excimer Laser Surface Ablation in Combination With Corneal Cross-linking (CCL) in Patients With Progressive Ectatic Corneal Disorders.
Brief Title: Corneal Cross Linking and Topography Guided Excimer Laser Treatment
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerald Schmidinger, MD, Assistant Professor, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 367/2009
Record Dates: First submitted 2011-11-05; First posted 2012-09-11 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Keratoconus; Pellucid Marginal Degeneration
Keywords: corneal cross linking; topography guided excimer laser; Keratoconus; Pellucid marginal degeneration; Post Excimer ectasia
MeSH Terms: conditions — Keratoconus | interventions — Corneal Cross-Linking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Corneal Cross Linking (Active Comparator): Patients will receive a standard corneal cross linking treatment
  Interventions: Other: Corneal Cross Linking
- Corneal Cross Linking and Topo Laser (Experimental): Patients will receive a topography guided laser treatment in combination with a standard corneal cross linking treatment in the same session.
  Interventions: Other: Topography guided Excimer Laser treatment and Corneal Cross Linking

INTERVENTIONS:
Other: Topography guided Excimer Laser treatment and Corneal Cross Linking — A topography guided excimer laser treatment will be performed prior to CCL in one session.
  Arms: Corneal Cross Linking and Topo Laser
Other: Corneal Cross Linking — A standard corneal cross linking procedure will be performed in this arm.
  Arms: Corneal Cross Linking

SUMMARY:
Topography guided laser treatment enables the surgeon to correct higher order aberrations in corneas with irregular astigmatism. Several case reports and small uncontrolled trials have been published on the combination of this treatment with corneal cross linking (CCL) in patients with ectatic corneal diseases.

This randomized study will evaluate the safety and efficacy of a combined treatment of corneal cross linking with a partial topography guided excimer laser treatment in eyes with progressive ectatic corneal diseases.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Patient age 18 - 40 years
* Documented progressive corneal ectatic disease except post LASIK/LASEK ectasia

Exclusion Criteria:

* Allergy to one of the used substances
* Tendency towards excessive scar formation
* Pregnancy
* Rheumatic diseases
* Central corneal thickness below 450 µm
* Active infection of the study eye
* Previous corneal surgery of the study eye

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Safety (Pachymetry, K-readings) | 1 year
uncorrected visual acuity (UVCA) | 1 year
best corrected visual acuity (BCVA) | 1 year

SECONDARY OUTCOMES:
Progression of ectatic disease (by use of maximum keratometry readings = Kmax) | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Department of Ophthalmology, Vienna, Austria